CLINICAL TRIAL: NCT00054626
Title: Phase III Study Of Adjuvant Cisplatin-Gemcitabine Vs. Observation After Radical Cystectomy In High-Risk Bladder Cancer
Brief Title: Cisplatin and Gemcitabine Compared With Observation in Treating Patients Who Have Undergone Surgery for Bladder Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000258426; ITNRC-CU02.00447ST/97; NCI-V02-1715
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2008-11

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known if combination chemotherapy is effective in preventing relapse in patients who have undergone radical cystectomy for bladder cancer.

PURPOSE: Phase III trial to compare the effectiveness of cisplatin combined with gemcitabine with that of observation in treating patients with bladder cancer who have undergone surgery to remove the bladder.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall, cause-specific, and disease-free survival of patients with high-risk muscle-invasive transitional cell carcinoma of the bladder treated with adjuvant cisplatin and gemcitabine vs observation after radical cystectomy.
* Compare the dose intensity and toxicity of two different schedules of cisplatin and gemcitabine in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and disease status (T2 [G3 only] or T3-4 [any G], N0-2 vs any T, N1-2, M0). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients are further randomized to 1 of 2 treatment regimens.

  * Regimen A: Patients receive cisplatin IV on day 2 and gemcitabine IV on days 1, 8, and 15.
  * Regimen B: Patients receive cisplatin IV on day 15 and gemcitabine as in regimen A.

Treatment in both regimens repeats every 28 days for 4 courses.

* Arm II: Patients undergo observation followed by cisplatin and gemcitabine as in arm I at relapse.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 700 patients (350 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the bladder

  * T2 (G3 only) or T3-4 (any G), N0-2 or any T, N1-2, M0
  * No secondary localization
* Radical cystectomy (without residual disease) performed within 10 weeks prior to study entry to include:

  * Men: Cystectomy with removal of prostate and seminal vesicles including 1.5 cm of urethra plus pelvic lymphadenectomy (at least 15 negative lymph nodes are recommended to define as N0)
  * Women: Cystectomy with complete removal of the bladder, uterus, ovaries, and anterior walls of the vagina plus pelvic lymphadenectomy

PATIENT CHARACTERISTICS:

Age

* 18 to 74

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,500/mm^3
* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin less than upper normal limit (ULN)
* Gamma-GT less than ULN
* SGOT and SGPT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal

* Creatinine no greater than1.25 times ULN
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No congestive heart failure
* No angina pectoris
* No cardiac arrhythmia
* No uncontrolled arterial hypertension
* No history of acute myocardial infarction within the past year

Other

* No other serious concurrent illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Palliative radiotherapy allowed at relapse for symptomatic bone metastases

Surgery

* See Disease Characteristics

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2001-09; Primary Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 5 years

SECONDARY OUTCOMES:
Disease-free survival at 5 years
Local disease-free survival at 5 years
Distant disease-free survival at 5 years
Toxicity by WHO system grading after each course
Quality of life after each course and every 6 months during follow-up
Dose intensity at the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Camillo F. Pollera, MD, Study Chair — Presidio Ospedaliero Belcolle
Locations (151):
- Italy (151):
  - Ospedale Civile Via Caronia, Acireale - CT
  - Ospedale San Lazzaro, Alba
  - Ospedale S. Giuseppe, Albano Laziale
  - Ospedale SS. Biagio e Arrigo, Alessandria
  - Ospedale Civile Alessandria, Alessandria
  - Presidio Ospedale, Anagni
  - Ospedale Torrette University Ancona, Ancona
  - Ospedale Generale Umberto 1, Ancona
  - Istituto Nazionale Riposo e Cura Anziani Istituto, Ancona - AN
  - Ospedale S. Donato, Arezzo
  - Ospedale Civile di Asti, Asti
  - S.G. Moscati Hospital, Avellino
  - Ospedale Civile Avezzano, Avezzano
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Universita Degli Studi di Bari, Bari
  - Istituto Di Ricovero E Cura A Carattere Scientifico, Bari
  - Ospedale di Venere - Carbonara, Bari-Carbonara
  - Ospedale S. Martino, Belluno
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale degli Infermi - ASL 12, Biella
  - Azienda Ospedaliera Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Sanitaria di Bolzano, Bolzano
  - Ospedale S. Trinita, Borgomanero
  - Spedali Civili di Brescia, Brescia
  - Ospedale di Busto Arsizio, Busto Arsizio
  - Ospedale SS Trinita, Cagliari
  - Ospedale Caltanissetta, Caltanissetta
  - Ospedale Civile Camposanpiero, Camposanpiero
  - Istituto per la Ricerca e Cura del Cancro, Candiolo
  - Civic Hospital of Carrara, Carrara
  - Ospedale S. Spirito, Casale Monferrato
  - Ospedale S. Leonardo, Castellammare Di Stabia - NA
  - Ospedale Cannnizzaro, Catania
  - Ospedale S. Luigi, Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Ospedale SS Annunziata, Chieti
  - Universita G.D'Annunzio Di Chieti, Chieti
  - Ospedale Di Cirie, Cirié
  - Ospedale Sant Anna, Como
  - Ospedale Maggiore Crema, Crema
  - Ospedale Civile S. Croce, Fano
  - Ospedale Fidenza, Fidenza
  - Ospendale S.M. Annunziata-A.S.DI Florence, Florence
  - Morgagni-Pierantoni Ospedale, Forlì
  - Ospedale S. Sebastiano, Frascati - RM
  - Ospedale Umberto I, Frosinone
  - Ospedale S. Antonio Abate, Gallarate Varese
  - Ospedale Di Gela, Gela - CL
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Ospedale San Martino, Genoa
  - Presidio Ospedaliero-Gorizia, Gorizia
  - Ospedale Misericordia USL 9, Grosseto
  - INI Grottaferrata, Grottaferrata
  - Ospedale Nuovo, Imola
  - Ospedali Vecchi, Imola
  - Ospedale Civile di Ivrea, Ivrea
  - Ospendale S. Andrea EST, La Spezia
  - Ospedale Civile Lanciano, Lanciano
  - Ospedale Santa Maria Goretti, Latina
  - Ospedale Alessandro Manzoni, Lecco
  - Ospedale Civile di Legnano, Legnano
  - Presidio Ospedaliero di Livorno, Livorno
  - Carlo Poma Hospital, Mantova
  - Ospedale Papardo, Messina
  - Policlinico Messina, Messina
  - University of Milan, Milan
  - Ospedale San Giuseppe, Milan
  - Istituto Scientifico H. San Raffaele, Milan
  - European Institute of Oncology, Milan
  - Ospedale Fatebene Fratelli, Milan
  - Ospedale San Carlo Borromeo, Milan
  - Ospedale Luigi Sacco, Milan
  - Azienda Ospedaliera - Universitaria di Modena, Modena
  - Sant Agostino - Estenes Institutes, Modena
  - Policlinico Monserrato, Monserrato - CA
  - Clinica Urologica II, Monza
  - Ospedale San Gerardo, Monza
  - Azienda Ospedaliera "A. Cardarelli", Naples
  - Federico II University Medical School, Naples
  - Istituto Tumori/Fondazione Pascale, Naples
  - Ospedale Civile Negrar, Negrar
  - Azienda Ospedaliera Maggiore Della Carita, Novara
  - Azienda Ospedale S. Luigi at University of Torino, Orbassano
  - Casa di Cura Noto Pasqualino, Palermo
  - Ospedale Oncology M. Ascoli, Palermo
  - Ospedale La Maddalena - Palermo, Palermo
  - Azienda Ospedaliera Di Parma, Parma
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Universita Degli Studi, Pavia
  - Azienda Ospedale - d "S. Salvatore", Pesaro
  - Ospedale Spiritito Santo, Pescara
  - Ospedale Santa Corona, Pietra Ligure -SV
  - Ospedale Santa Chiara Pisa, Pisa
  - Ospedale Pistoia, Pistoia
  - Azienda Ospedaliera "Santa Maria Degli Angeli", Pordenone
  - Azienda U.S.L. Cesena, Potenza
  - Ospedale Carlo Forlanini, Potenza
  - Ospedale Di Rivoli, Rivoli
  - Azienda Ospedaliera Sant'Andrea, Rome
  - Ospedale C.T.O. Roma, Rome
  - Ospedale Sant' Eugenio, Rome
  - Azienda Ospedaliera S. Camillo-Forlanini, Rome
  - Azienda Policlinico Umberto Primo, Rome
  - Istituto Regina Elena, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Fatebenefratelli, Isola Tiberina Hospital, Rome
  - Ospedale San Pietro Fatebenefratelli, Rome
  - Ospedale Civile di Rovigo, Rovigo
  - Istituto Clinico Humanitas, Rozzano
  - Ospedale Saluzzo, Saluzzo - CN
  - Ospedale San Daniele del Friuli, San Daniele del Friuli
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale Civile Di San Vito Al Tagliamento, San Vito Al Talgliamento
  - Az. Ospedale Villa Scassi, Sandpierdarena
  - ASL NO. 1 Imperiese, Sanremo
  - Ospedale Civile G Borea, Sanremo
  - Istituto Clinica Medica, Sassari
  - Ospedale Civile ASL 1, Sassari
  - Ospedale SS Trinita, Sassari
  - Policlinico Sassari, Sassari
  - Ospedali Savigliano, Savigliano - CN
  - Ospedale S. Paolo Valloria, Savona
  - Ospedale Civile Sestri Levante, Sestri Levante - GE
  - Universita di Siena, Siena
  - Osepdale Civile, Sondrio
  - Ospedale SS Trinita, Sora
  - SS Annunziata, Sulmona
  - Ospedale Umberto 1, Syracuse
  - Ospedale S. Vincenzo, Taormina
  - Ospedale Civile Teramo, Teramo
  - Ospedale Generale Prov. Boldrini, Thiene
  - Ospedale Civile, Tolmezzo Gemona F.
  - Ospedale Civile Trapani, Trapani
  - Ospedale Di Trento, Trento
  - Primario U.O. di Oncologia Medica, Trento
  - Ospedale Cattinara, Trieste
  - Ospedale Amedeo Savoia, Turin
  - Ospedale Martini, Turin
  - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Turin
  - Ospedale Gradenigo, Turin
  - Ospedale Cottolengo, Turin
  - Ospedale Giovanni Bosco, Turin
  - Ospedale S. Giovanni Vecchio, Turin
  - Azienda Ospedaliera Santa Maria della Misericordia, Udine
  - Ospedale Civile ULSS 12, Venezia
  - Ospedale Civile Verbania, Verbania
  - Ospedal San Andrea, Vercelli
  - Policlinico Borgo Roma, Verona
  - Policlinico G. B. Rossi - Borgo Roma, Verona
  - Ospedale San Bortolo, Vicenza
  - Presidio Ospedaliero Belcolle, Viterbo

REFERENCES:
- [Result] Pollera CF, Merendino N, Cianciulli AM, et al.: Preliminary cytogenetic and pharmacogenomic analysis of muscle-invasive transitional-cell carcinoma (TCC) of the bladder in patients (pts) enrolled in the Italian National Research Council (CNR) phase III randomized trial comparing adjuvant cisplatin-gemcitabine (PG) vs observation (OBS) after radical cystectomy. [Abstract] J Clin Oncol 23 (Suppl 16): A-4589, 400s, 2005.